CLINICAL TRIAL: NCT01533285
Title: A 2-way Crossover Study to Explore the Effect of an Inflammatory and Psychosocial Stressor and a Combination Thereof on the Mood and Cytokine Levels in Young and Elderly Healthy Female Subjects and Female Subjects With Major Depressive Disorder
Brief Title: Exploratory Study on the Mood and Cytokine Levels in Female Healthy Participants and Major Depressive Disorder Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: CR100698; NOCOMPOUNDEDI0002 (Other: Janssen Pharmaceutica N.V.); 2011-004898-80 (EudraCT Number)
Record Dates: First submitted 2012-01-19; First posted 2012-02-15 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Major Depressive Disorder
Keywords: Major depressive disorder; MDD; Psychiatry disorders; Psychosocial stressor; Psychosocial stress; Typhoid vaccination; Typhoid vaccine
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Vi polysaccharide vaccine, typhoid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Group 1 (Other): Treatment AB: Treatment A (Placebo vaccination) administered [Period 1], after the washout period (7-14 days) Treatment B (typhoid vaccination) administered [Period 2]
  Interventions: Biological: Placebo; Biological: Salmonella typhi vaccine (Typhim Vi)
- Group 2 (Other): Treatment BA: Treatment B (typhoid vaccination) administered [Period 1], after the washout period (7-14 days) Treatment A (Placebo vaccination) administered [Period 2]
  Interventions: Biological: Placebo; Biological: Salmonella typhi vaccine (Typhim Vi)
- Group 3 (Other): Treatment AC: Treatment A (Placebo vaccination) administered [Period 1], after the washout period (7-14 days) Treatment C (TSST+Placebo vaccination) administered [Period 2]
  Interventions: Biological: Placebo
- Group 4 (Other): Treatment CA: Treatment C (TSST+Placebo vaccination) administered [Period 1], after the washout period (7-14 days) Treatment A (Placebo vaccination) administered [Period 2]
  Interventions: Biological: Placebo
- Group 5 (Other): Treatment AD:Treatment A (Placebo vaccination) administered [Period 1], after the washout period (7-14 days) Treatment D (TSST+typhoid vaccination) administered [Period 2]
  Interventions: Biological: Placebo; Biological: Salmonella typhi vaccine (Typhim Vi)
- Group 6 (Other): Treatment DA:Treatment D (TSST+typhoid vaccination) administered [Period 1], after the washout period (7-14 days) Treatment A (Placebo vaccination) administered [Period 2]
  Interventions: Biological: Placebo; Biological: Salmonella typhi vaccine (Typhim Vi)

INTERVENTIONS:
Biological: Placebo — Placebo is Treatment A and C. Form=saline solution for intramuscular (IM) injection (Injection of a solution into a muscle), route = IM, Unit = mL, number = 0.5 administered on Day 1 of Period 1 and Period 2.
Biological: Salmonella typhi vaccine (Typhim Vi) — Salmonella typhi vaccine (typhoid vaccination) in Treatment B and D; Unit = mg, number = 0.025, form = solution for intramuscularly (IM) injection, route = IM administered on Day 1 of Period 1 and Period 2.
  Arms: Group 1; Group 2; Group 5; Group 6

SUMMARY:
The purpose of this study is to explore the effect of an inflammatory and a psychosocial stressor and the combination thereof on mood in healthy young and elderly participants and patients with Major Depressive Disorder (MDD).

DETAILED DESCRIPTION:
This is a 2-way crossover (method used to switch patients from one treatment arm to another in a clinical study), randomized (the study medication is assigned by chance), placebo-controlled (an inactive substance that is compared with a study medication to test whether the medication has a real effect in a clinical study) study in 3 cohorts (group of individuals with similar characteristics) ie, 18 healthy young female participants; 18 healthy elderly female participants; 18 female patients with a past history of MDD. Participants will be randomized to 1 of 6 possible treatment groups: Group 1: Treatment AB, Group 2: Treatment BA, Group 3: Treatment AC, Group 4: Treatment CA, Group 5: Treatment AD, Group 6: Treatment DA, where Treatment A is placebo vaccination, Treatment B is typhoid vaccination, Treatment C is psychosocial stress (Trier Social Stress Test [TSST]) followed by placebo vaccination, and Treatment D is psychosocial stress (TSST) followed by typhoid vaccination. Participants from each of the 3 cohorts will be randomized to these 6 treatment groups. In all the 6 groups the 1st treatment comes under Period 1 and 2nd treatment under Period 2 (eg, In Group 1: Treatment A [Period 1] and Treatment B [Period 2]) and there will be a minimally 7- and maximally 14- day washout period (period when no treatment is received) between the study periods. The study will consist of an eligibility screening examination (from 21 to 2 days prior to Day 1 of Period 1); a run-in visit (only prior to Period 1) in which eligible participants will be briefly explained about the cognitive test battery and immediately thereafter the baseline of cognitive function will be measured via these tests; 2 single-blind (a clinical study in which the person giving the treatment, but not the patient, knows which treatment the patient is receiving) treatment periods (2-way crossover); and a follow-up examination by phone (approximately 7 to 14 days after last treatment [Period 2]). For each participant, the maximal study duration will not exceed 8 weeks.

ELIGIBILITY:
Inclusion criteria:

* Has body mass index (BMI) [weight in kilograms / (height in meters x height in meters)] between 18 and 30 kg/m2
* For young healthy participants: female, 25 to 45 years of age; elderly healthy participants: female: ≥ 65 years of age & with baseline C-reactive protein (CRP) > 5 mg/mL; (partially) remitted MDD patients: female, 25 to 45 years of age
* Inclusion criteria specific for patients with MDD: -Patients with a history (within 24 months) of MDD must have a Montgomery-Asberg Depression Rating Scale (MADRS) total score < 15 and symptom remission (temporary absence of disease symptoms) relative to the acute episode must have been present for at least 3 months

Exclusion Criteria:

* Has a current Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) axis I diagnosis (other than MDD)
* Has recently experienced a psychosocial stressor within 6 months
* Has acute symptoms of suicidality (the likelihood of an individual completing suicide)
* Has a DSM-IV diagnosis of substance abuse or dependence within 6 months prior to screening evaluation
* Has been exposed to an experimental medication or experimental medical device within 90 days before screening
* Has a serology (scientific study of blood serum and other bodily fluids) positive for hepatitis B surface antigen (HBsAg), hepatitis C antibodies or HIV antibodies at screening
* Has been exposed to typhoid or typhoid vaccine within 5 years before screening
* Has been prior exposed to the Trier Social Stress Test (TSST)
* Has received electroconvulsive therapy (shock therapy) within 3 months before screening
* Has been involuntarily committed to psychiatric hospitalization
* Has donated 1 or more units (approximately 450 mL) of blood or had an acute loss of an equivalent amount of blood within 90 days prior to study medication administration

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-05; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Change in Profile of Mood States (POMS) scores from Baseline to Day 1 of Period 1 and Period 2. | Baseline (pretreatment), Day 1 of Period 1 and Period 2.
  Participants score on a scale ranging from 0 (not at all) to 4 (extremely) any of 30 statements related to their mood / energy level by circling the appropriate number.
Change in Visual Analogue Scale (VAS) scores from Baseline to Day 1 of Period 1 and Period 2. | Baseline (pretreatment), Day 1 of Period 1 and Period 2.
  Participants rate the way they feel on a 10 mm line separating statements along the extremes of different dimensions (eg, alert - drowsy).
Change in Snaith-Hamilton Pleasure Scale (SHAPS) scores from Baseline to Day 1 of Period 1 and Period 2. | Baseline (pretreatment), Day 1 of Period 1 and Period 2.
  Participants endorse any of 14 statements in 4 categories (Strongly Agree, Agree, Disagree, Strongly Disagree) by ticking the appropriate answer.
Change in Montgomery-Asberg Depression Rating Scale (MADRS) scores from Baseline to Day 1 of Period 1 and Period 2. | Baseline (pretreatment), Day 1 of Period 1 and Period 2.
  The MADRS is used by trained blinded site staff to rate the severity of depression. It consists of 10 items. The minimal rating is 0 (absent) and the maximal rating is 6 (most serious).

SECONDARY OUTCOMES:
Change in Cognitive Test Battery performance from Baseline to Day 1 of Period 1 and Period 2. | Baseline (≤ Day -1 [1 day before starting study drug]), Day 1 of Period 1 and Period 2.
  Performance in cognitive tests after the inflammatory (vaccination) and psychosocial stressor and the combination thereof. The cognitive domains to be tested include attention, emotional bias, memory, and executive functioning.
Changes in levels of hormones and cytokines from Baseline to Day 1 of Period 1 and Period 2. | Baseline (pretreatment), Day 1 of Period 1 and Period 2.
  Changes in levels of hormones and cytokines after the inflammatory (vaccination) and psychosocial stressor and the combination thereof. Approximately 10 mL of blood samples from veins must be collected for the assessment of hormones and cytokines (protein released by cells in blood) related to inflammation and depression (or other relevant neuropsychiatric disorders).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V. Clinical Trial, Study Director — Janssen Pharmaceutica N.V.
Locations (2):
- Belgium (2):
  - Duffel
  - Leuven

REFERENCES:
- [Derived] Niemegeers P, de Boer P, Schuermans J, Dumont GJH, Coppens V, Spittaels K, Claes S, Sabbe BGC, Morrens M. Digging deeper in the differential effects of inflammatory and psychosocial stressors in remitted depression: Effects on cognitive functioning. J Affect Disord. 2019 Feb 15;245:356-363. doi: 10.1016/j.jad.2018.11.020. Epub 2018 Nov 6. PMID 30423462